CLINICAL TRIAL: NCT00002819
Title: A RANDOMIZED, CONTROLLED TRIAL OF SALVAGE THERAPY WITH PACLITAXEL AND CARBOPLATIN VERSU SALVAGE THERAPY WITH STEM CELL SUPPORTED HIGH-DOSE CARBOPLATIN, MITOXANTRONE AND CYCLOPHOSPHAMIDE IN PATIENTS WITH PERSISTENT LOW VOLUME OVARIAN CANCER AND RESPONSE TO PRIMARY THERAPY
Brief Title: Chemotherapy With or Without Peripheral Stem Cell Transplantation in Treating Patients With Persistent Ovarian Epithelial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064983; GOG-164; CLB-9791; E-G0164; SWOG-G0164
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2007-05

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Cyclophosphamide; Mitoxantrone; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: mitoxantrone hydrochloride
Drug: paclitaxel
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. It is not yet known whether chemotherapy alone is more effective than chemotherapy plus peripheral stem cell transplantation for ovarian epithelial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel and carboplatin with that of carboplatin, mitoxantrone, and cyclophosphamide followed by peripheral stem cell transplantation in treating patients who have persistent stage III or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare progression-free and overall survival of patients with drug-sensitive, low-volume ovarian cancer that is persistent following standard therapy treated with salvage therapy comprising standard-dose paclitaxel and carboplatin vs high-dose carboplatin, mitoxantrone, and cyclophosphamide followed by bone marrow reconstitution. II. Compare the toxic effects of these two salvage regimens. III. Compare selected health-related aspects of quality of life in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating center and disease state at reassessment laparotomy. Patients are randomized to one of two treatment arms. Arm I: Patients receive paclitaxel IV over 3 hours on day 1 and carboplatin IV continuously on days 1-5 every 3 weeks for a total of 6 courses. Arm II: Patients receive cyclophosphamide IV over 1 hour and mitoxantrone IV over 15 minutes on days -8, -6, and -4, and carboplatin IV continuously on days -8 through -4, followed by rescue with autologous bone marrow or peripheral blood stem cells on day 0. Quality of life is assessed at baseline, at 3 and 9 weeks after starting treatment, and every 3 months for an additional 5 assessments regardless of disease progression.

PROJECTED ACCRUAL: A total of 275 patients will be accrued over approximately 60 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV ovarian epithelial carcinoma including the following cellular diagnoses: Serous adenocarcinoma Mucinous adenocarcinoma Endometrioid adenocarcinoma Clear cell adenocarcinoma Undifferentiated carcinoma Mixed epithelial carcinoma Transitional cell carcinoma Malignant Brenner's Tumor Stage III (optimal or suboptimal) must be surgically reassessed OR Stage III (suboptimal) or stage IV clinically reassessed after induction chemotherapy For stage III surgical reassessment: No more than 12 weeks between end of chemotherapy and reassessment surgery AND No more than 6 weeks between reassessment surgery and randomization Patients treated on protocol GOG-158 are eligible At least a partial response to chemotherapy as defined as: Microscopic disease documented at reassessment surgery for patients optimally debulked (disease no greater than 1 cm) after primary surgery Suboptimally debulked disease (greater than 1 cm) after primary surgery and 1 of the following: Negative reassessment laparotomy Only microscopic disease at reassessment surgery Gross residual disease no greater than 1 cm at reassessment surgery prior to debulking Clinical complete response to induction chemotherapy including: - suboptimal disease Stage III or IV AND - either an abnormal CT or elevated CA-125 prior to induction chemotherapy and both are within normal limits following induction chemotherapy

PATIENT CHARACTERISTICS: Age: Under 66 Performance status: GOG 0 or 1 Hematopoietic: Absolute granulocyte count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 3 times normal Renal: Creatinine clearance at least 60 mL/min Cardiovascular: Left ventricular ejection fraction at least 45% by MUGA No congestive heart failure Pulmonary: FEV1 and FVC at least 60% Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No prior malignancy in the past 5 years except adequately treated nonmelanomatous skin cancer, carcinoma in situ of the cervix, or any other cancer whose prior treatment does not contraindicate this study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 and no more than 6 prior platinum-based combination chemotherapy courses (i.e., cisplatin or carboplatin) required Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No prior anthracyclines

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-11; Primary Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P. McGuire, MD, Study Chair — Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center; Kenneth B. Miller, MD, Study Chair — Tufts Medical Center Cancer Center; Patrick J. Stiff, MD, Study Chair — Loyola University; Stephen L. Graziano, MD, Study Chair — State University of New York - Upstate Medical University
Locations (64):
- United States (64):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin